CLINICAL TRIAL: NCT04455347
Title: Cardiac and Thoracic Imaging in Pediatric Patients With Evidence of Systemic Inflammation COVID19 Linked
Acronym: CARDOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HJ-20-CARDOVID
Record Dates: First submitted 2020-07-01; First posted 2020-07-02 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Infection
Keywords: COVID-19 Infection; Children; Acute Myocarditis; Kawasaki-like-syndrome
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To perform comprehensive cardiac and thoracic non invasive imaging assessment by MRI and/or CT scan including cardiac functional evaluation and myocardial tissue characterization of COVID_19 related disease in pediatric patients with cardiac involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with cardiac MRI or cardiac CT scan or thoracic CT scan admitted for acute inflammatory syndrome and cardiac compromise
2. Patient with PCR or antibodies test for COVID 19 (positive of negative)
3. Patient or parents of minor patients informed about collection of personal data for the study

Exclusion Criteria:

* Patient or parents refusing personal data collection

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with a probable or a proven diagnosis of COVID 19 admitted for systemic acute inflammation and cardiac symptoms (cardiogenic shock or chest pain or clinical suspicion of acute myocarditis or left ventricular ejection fraction)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Imaging data at Baseline | Baseline
  Description of imaging data from MRI ans CT scan and associated clinical data.
Imagine data at Follow-up | During the 2 years follow-up period
  Description of imaging data from MRI ans CT scan and associated clinical data.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Raimondi, MD, Principal Investigator — Hôpital Necker
Locations (1):
- Hôpital Necker, Paris, France

REFERENCES:
- [Derived] Aeschlimann FA, Misra N, Hussein T, Panaioli E, Soslow JH, Crum K, Steele JM, Huber S, Marcora S, Brambilla P, Jain S, Navallas M, Giuli V, Rucker B, Angst F, Patel MD, Azarine A, Caro-Dominguez P, Cavaliere A, Di Salvo G, Ferroni F, Agnoletti G, Bonnemains L, Martins D, Boddaert N, Wong J, Pushparajah K, Raimondi F. Myocardial involvement in children with post-COVID multisystem inflammatory syndrome: a cardiovascular magnetic resonance based multicenter international study-the CARDOVID registry. J Cardiovasc Magn Reson. 2021 Dec 30;23(1):140. doi: 10.1186/s12968-021-00841-1. PMID 34969397